CLINICAL TRIAL: NCT00175461
Title: Comparison of the Clinical Effectiveness and Cost-effectiveness of the MIS Anterolateral Approach (MIS Watson Jones, G3) Versus Anterolateral Mini or Posterolateral Mini Approaches in Primary Total Hip Arthroplasty
Brief Title: Comparison of Two Minimally Invasive Surgical Techniques for Hip Replacement
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of British Columbia (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: H04-70070
Record Dates: First submitted 2005-09-11; First posted 2005-09-15 (Estimated); Last update posted 2017-03-03 (Actual); Status verified 2017-03

CONDITIONS: Osteoarthritis
MeSH Terms: conditions — Osteoarthritis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Procedure: hip surgery — Comparison of the clinical effectiveness and cost-effectiveness of the MIS anterolateral approach (MIS Watson Jones, G3) versus anterolateral mini or posterolateral mini approaches in primary total hip arthroplasty

SUMMARY:
Comparison of the clinical effectiveness and cost-effectiveness of the MIS anterolateral approach (MIS Watson Jones, G3) versus anterolateral mini or posterolateral mini approaches in primary total hip arthroplasty

ELIGIBILITY:
Inclusion Criteria:

No contralateral hip symptoms, no major comorbidity

Exclusion Criteria:

-

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 156 (Actual)
Dates: Start 2005-09; Primary Completion 2009-04 (Actual); Study Completion 2011-08-31 (Actual)

PRIMARY OUTCOMES:
3-months WOMAC score | 3 months

SECONDARY OUTCOMES:
Cost-effectiveness at 2-years | Two years

CONTACTS AND LOCATIONS:
Overall Officials: Nelson Greidanus, MD, Principal Investigator — University of British Columbia
Locations (1):
- Vancouver General Hospital, Vancouver, British Columbia, Canada